CLINICAL TRIAL: NCT01986725
Title: The Impact of the Self-management Intervention "WOMAN-PRO II Program" on Patients With Vulvar Neoplasia to Minimize Post-surgical Symptom Prevalence: A Mixed-Methods Project
Brief Title: The Impact of the "WOMAN-PRO II Program" on Patients With Vulvar Neoplasia to Minimize Post-surgical Symptom Prevalence
Acronym: WOMAN-PROII
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St.Gallen University of Applied Sciences (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other); University Hospital, Basel, Switzerland (Other); Cantonal Hospital of St. Gallen (Other); Medical University of Vienna (Other); Cantonal Hospital of Lucerne, Switzerland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: WOMAN-PRO II program
Record Dates: First submitted 2013-05-21; First posted 2013-11-18 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Vulvar Cancer; Vulvar Intraepithelial Neoplasia
Keywords: vulvar neoplasia; vulvar cancer; vulvar intraepithelial neoplasia; self management; symptom management
MeSH Terms: conditions — Vulvar Neoplasms | interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standardized care (Active Comparator): During treatment and routine follow-up consultations, patients randomized to standardized care will be provided with usual care and a predefined set of additional written information leaflets about supportive care options in the early treatment phase designed for the study.
  Interventions: Behavioral: standardized care (Intervention I)
- Standardized care + WOMAN-PRO II program (Active Comparator): During treatment and routine follow-up consultations, patients randomized to standardized care + WOMAN-PRO II program will be provided with usual care and nurse-led follow-up consultations with the WOMAN-PRO II program complementary to physician appointments.
  Interventions: Behavioral: Standardized care + WOMAN-PRO II program (Intervention II)

INTERVENTIONS:
Behavioral: standardized care (Intervention I) — During treatment and routine follow-up consultations, patients randomized to standard care will be provided with usual care and a predefined set of additional written information leaflets about supportive care options in the early treatment phase designed for the study.Usual care includes treatment during hospitalization by the gynecologist and the nurses according to the existing guidelines. At each follow-up visit, the gynecologist will conduct a physical examination. The follow-ups include also treatment of adverse effects of the therapy and rehabilitation.
  Arms: Standardized care
Behavioral: Standardized care + WOMAN-PRO II program (Intervention II) — This intervention is in addition to standard care. Nurse-led follow-up consultations with the WOMAN-PRO II program complementary to physician appointments have the goal to support women's self-management abilities in order to deal with occurring symptoms and related distress. Content of the WOMAN-PRO II program designed for this study is summarized in a handbook for professionals including patient clinical pathways and nurse interventions, supplemented by a patient booklet (paper based and electronic version) with tailored information according to patients' needs. The program includes five consultations with an approximate total duration of two hours.
  Arms: Standardized care + WOMAN-PRO II program

SUMMARY:
In vulvar neoplasia, even minor surgical interventions cause multiple symptoms, symptom distress and complications, which have an impact on a woman's quality of life and contribute to high health care costs. For the majority of the patients, symptom and distress can be reduced if adequate treatment is provided. This study aims to test possible differences between the impact of standardized care and the WOMAN-PRO II program on symptom prevalence in women with vulvar neoplasia after surgical treatment.

In a sequential explanatory mixed-methods project, a randomized phase II study will be followed by a qualitative sub-study. Ninety patients with vulvar neoplasia treated surgically will participate in the randomized trial in four Swiss hospitals and one Austrian hospital. After stratification by precancer/cancer, women will be randomly assigned (1:2 ratio) to standardized care and the WOMAN-PRO II program. The standardized care group will receive a set of information leaflets about supportive care options in the clinic. The WOMAN-PRO II program group will obtain counseling sessions by specially trained gynecology-oncology nurse specialists at the moment of diagnosis, 7 days post-surgery, in week two after discharge, week twelve and week 24 after surgery. The primary outcome of this study is symptom prevalence. Secondary outcomes will be collected for explorative reasons and include symptom distress, uncertainty, quality of life, social support, resilience, quality of care, sociodemographic and medical characteristics, post-surgical complications, functional status, cost evaluation and process outcomes. Quantitative data will be collected at the counseling points of time and analyzed by using mixed linear regression analysis. Twenty interviews will be conducted with women of the WOMAN-PRO II program group. A focus-group interview will be conducted with twelve gynecology-oncology nurse specialists in order to better understand to which degree the interventions meet individual needs as well as to identify remaining barriers and enablers for the implementation of symptom self-management. Qualitative data will be analyzed by using thematic analysis and a critical hermeneutic reflection.

This study will evaluate the impact of the WOMAN-PRO II program on symptom prevalence, patient-reported outcomes and clinical parameters, and inform the design of a possible phase III study on the clinical efficacy of the program.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of vulvar intraepithelial neoplasia (VIN) or vulvar cancer (primary diagnosis or recurrent neoplasia)
* Surgical treatment of VIN or vulvar cancer in one of the designated hospitals
* Age > 18

Exclusion Criteria:

* Patients being judged by a physician or by a gynecology-oncology nurse specialist as not being capable to participate in the trial and to complete the questionnaire due to cognitive, linguistic, emotionally or physically reasons.
* Patients in concurrently psychiatric treatment
* Terminal illness

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Changes in symptom prevalence | Change from baseline symptom prevalence at 6 months, measured on the following points of time: diagnosis, 7 days post-surgery, week two after discharge, week twelve and week 24 after surgery
  The primary endpoint of the quantitative study is symptom prevalence, defined as a number of occurring symptoms on predefined time points from diagnosis (t0) across repeated measurements to follow-up assessment at six months after surgery (t4) Symptom prevalence after surgical treatment of vulvar neoplasia will be measured with the German WOMAN-PRO symptom diary. This self-report patient-reported outcome measure covers 31 symptoms occurring after surgery: 15 wound-related symptoms, 5 difficulties in daily life and 11 items that inquire about psychosocial feelings, thoughts or activities. For wound-related symptoms and difficulties in daily life, women are asked to rate how frequently they experienced the symptom/difficulty during the last seven days (never, for 1-2 days, 3-4 days, or 5-7 days).

SECONDARY OUTCOMES:
Changes in symptom severity | Change from baseline symptom severity at 6 months.
  Symptom severity after surgical treatment of vulvar neoplasia will also be measured with the WOMAN-PRO symptom diary. This self-report patient-reported outcome measure covers 31 symptoms occurring after surgery: 15 wound-related symptoms, 5 difficulties in daily life and 11 items that inquire about psychosocial feelings, thoughts or activities. For the psychosocial symptoms/issues, women are asked to assess the severity of symptoms (not at all, a little bit, quite a bit, very much).
Changes in Uncertainty-Mishel Uncertainty in Illness Scale (MUIS) | Change from baseline uncertainty at 6 months.
  The Mishel Uncertainty in Illness Scale (MUIS) is a 30-item scale detecting uncertainty in symptomatology, diagnosis, treatment, relationship with caregivers, and planning for the future.
Changes in the Health-related quality of life | Change from baseline health-related quality of life at 6 months
  The validated German and English Short Form (SF-36) will be administered. It utilizes scale profile, 36 questions and a one-week recall period. It contains eight subscale scores: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Items are rated on a 3-6-point Likert scale.
Changes in the perceived social support | change form baseline perceived social support at 6 months
  The Multidimensional Scale of Perceived Social Support (MSPSS) is a 12-item scale designed to assess three aspects of perceived social support. The tree aspects comprise support from friends, family, and significant others.
Changes in Resilience | Change from baseline reslilience at 6 months
  Resilience refers to positive adaptation following stress or trauma. The original Connor-Davidson Resilience Scale brief version (CD-RISC 10) is a 10-item scale assessing resilience during the last month, with higher scores indicating higher resilience capacity.
Changes in Patient Assessment of Chronic Illness Care | change from baseline Patient Assessment of Chronic Illness Care at 6 months
  The Patient Assessment of Chronic Illness Care (PACIC) instrument evaluates the quality and patient-centeredness of chronic illness care based on the Chronic Care Model (CCM)
Socio-demographic outcomes | baseline
  Socio-demographic outcomes for patients will be collected with an 11-items form concerning age, marital status, number of children, education, employment status, living situation, post surgical wound management at home, and health insurance. The instrument was developed for patients following vulvar surgical treatment.
Changes in clinical outcomes | change from baseline clinical outcomes at 6 months
  Clinical outcomes for patients will be collected with a 16-items form concerning diagnosis, cancer stage, initial treatment, and wound treatment. The instrument was developed for patients following vulvar surgical treatment.
Changes in functional status | Change from baseline functional status at 6 months.
  The functional status, referring to the capacity to perform a variety of activities that are normal for most people, will be measured with the Eastern Cooperative Oncology Group Performance Status (ECOG-PS). ECOG-PS is a one item five-point scale using verbal descriptors, ranging from 0 "fully active" to 5 "dead". It was developed in 1960 for cancer patients and has been widely used by physicians and researchers to assess how a patient's disease is progressing and how it affects the daily living abilities.
Changes in Assessment of Chronic Illness Care | Change from baseline assessment of chronic illness care at 6 months.
  The Assessment of Chronic Illness Care (ACIC) questionnaire was developed to assess if provided care is in alignment with the Chronic Care Model (CCM). The CCM comprises six areas: the organization of the health care system, the community linkage, self-management, decision support, delivery system design, and the clinical information system. The ACIC addresses how well a practice team or organization integrates the Chronic Care Model elements. Responses can be related to four descriptive levels from A "fully implemented" to D "little or none" implementation of the intervention.
Process outcomes | 6 months (baseline - 24 weeks following surgery)
  The collection of three process outcomes during the implementation of a complex intervention program will allow to draw conclusions about potential barriers and facilitators of the interaction between patient and gynecology-oncology nurse specialist during the counseling intervention. (1) Counseling competencies and details of the complex interaction between patients and the gynecology-oncology nurse specialist will be assessed during the study period by audio-recording a random sample of 15-20 counseling sessions.(2) The gynecology-oncology nurse will document her experiences after each counseling session by keeping a diary to reveal her personal situation during the counseling process. (3) The WOMAN-PRO II program teacher will contact the gynecology-oncology nurse specialists every eight weeks and document the content of the discussions by keeping a diary after each contact.
economic evaluation | 6 months (baseline - 24 weeks following surgery)
  Economic evaluation methods will be performed according to the recommendations of the NICE Reference Case. The economic evaluation will consist of a within-trial analysis and will compare direct costs and six-month outcomes of patients randomized to intervention II versus intervention I. Direct hospital costs will be the primary perspective. The study will record length of hospital stay, primary surgery costs, readmission, costs concerning intervention I, costs concerning intervention II, follow-up costs, patients non-productive time, and mortality. Comparison will be made between baseline and follow-up to estimate incremental cost-effectiveness ratio (ICER) comparing intervention II group with intervention I group in terms of the primary outcome measure (symptom prevalence) and costs.

CONTACTS AND LOCATIONS:
Overall Officials: Beate Senn, PhD, RN, Principal Investigator — Institute for Applied Nursing Sciences IPW, University of Applied Sciences FHS St. Gallen, Switzerland
Locations (1):
- Institute for Applied Nursing Sciences IPW, University of Applied Sciences FHS St. Gallen, Switzerland, Sankt Gallen, Switzerland

REFERENCES:
- [Result] Senn B, Eicher M, Mueller MD, Hornung R, Fink D, Baessler K, Hampl M, Denhaerynck K, Spirig R, Engberg S. A patient-reported outcome measure to identify occurrence and distress of post-surgery symptoms of WOMen with vulvAr Neoplasia (WOMAN-PRO) - a cross sectional study. Gynecol Oncol. 2013 Apr;129(1):234-40. doi: 10.1016/j.ygyno.2012.12.038. Epub 2013 Jan 3. PMID 23290987
- [Result] Senn B, Mueller MD, Cignacco EL, Eicher M. Period prevalence and risk factors for postoperative short-term wound complications in vulvar cancer: a cross-sectional study. Int J Gynecol Cancer. 2010 May;20(4):646-54. doi: 10.1111/IGC.0b013e3181d92723. PMID 20686386
- [Result] Senn B, Eicher M, Mueller MD, Engberg S, Spirig R. [Needs based nursing care in gynecology. "My symptom diary"]. Krankenpfl Soins Infirm. 2012;105(5):32-3. No abstract available. German. PMID 22675922
- [Result] Senn B, Mueller MD, Hasenburg A, Blankenstein T, Kammermann B, Hartmann A, Donovan H, Eicher M, Spirig R, Engberg S. Development of a postsurgical patient-reported outcome instrument for women with vulvar neoplasia. Oncol Nurs Forum. 2012 Nov;39(6):E489-98. doi: 10.1188/12.ONF.E489-E498. PMID 23107862
- [Result] Senn B, Eicher M, Mueller MD, Gafner D, Engberg S, Spirig R. [Development and validation of a patient reported outcome instrument for women with vulvar cancers and surgical treatment - a mixed method study]. Pflege. 2013 Feb;26(1):65-8. doi: 10.1024/1012-5302/a000265. No abstract available. German. PMID 23384847
- [Result] Gafner D, Eicher M, Spirig R, Senn B. [Between anxiety and hope: the experiences of women with vulval intraepithelial neoplasia during their illness trajectory - a qualitative approach]. Pflege. 2013 Apr;26(2):85-95. doi: 10.1024/1012-5302/a000273. German. PMID 23535473
- [Derived] Kofler S, Kobleder A, Ott S, Senn B. The effect of written information and counselling by an advanced practice nurse on resilience in women with vulvar neoplasia six months after surgical treatment and the influence of social support, recurrence, and age: a secondary analysis of a multicenter randomized controlled trial, WOMAN-PRO II. BMC Womens Health. 2020 May 6;20(1):95. doi: 10.1186/s12905-020-00965-z. PMID 32375773
- [Derived] Gehrig L, Kobleder A, Werner B, Denhaerynck K, Senn B. [Are written information or counseling (WOMAN-PRO II program) able to improve patient satisfaction and the delivery of health care of women with vulvar neoplasms? Secondary outcomes of a multicenter randomized controlled trial]. Pflege. 2017;30(5):257-269. doi: 10.1024/1012-5302/a000558. Epub 2017 Jun 27. German. PMID 28653559
- [Derived] Kobleder A, Raphaelis S, Glaus A, Fliedner M, Mueller MD, Gafner D, Gehrig L, Senn B. Recommendations for symptom management in women with vulvar neoplasms after surgical treatment: An evidence-based guideline. Eur J Oncol Nurs. 2016 Dec;25:68-76. doi: 10.1016/j.ejon.2016.10.003. Epub 2016 Oct 22. PMID 27865255